CLINICAL TRIAL: NCT05753202
Title: Neuromodulation Using Transcranial Direct Current Stimulation (tDCS) in Post-COVID Syndrome: Comparison of Two Targets
Brief Title: tDCS in Post-COVID Syndrome: Comparison of Two Targets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Jordi A Matias-Guiu, PhD MD, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22/728-P-EC
Record Dates: First submitted 2023-03-01; First posted 2023-03-03 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; Post-COVID-19 Syndrome; Post COVID-19 Condition
Keywords: post-COVID syndrome; brain stimulation; fatigue; cognitive; depression; transcranial direct current stimulation; non-invasive brain stimulation
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Fatigue; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left dorsolateral prefrontal cortex (Active Comparator): 15 sessiones of anodal tDCS over the left dorsolateral prefrontal cortex (2 mA, 20 minutes) associated with cognitive training.
  Interventions: Device: transcranial current direct stimulation
- Left M1 (Active Comparator): 15 sessiones of anodal tDCS over the left M1 (2 mA, 20 minutes) associated with cognitive training.
  Interventions: Device: transcranial current direct stimulation

INTERVENTIONS:
Device: transcranial current direct stimulation — Transcranial electrical stimulation over two different brain regions associated with cognitive training. 15 sesions in 3 weeks (5 days/week)

SUMMARY:
The main aim of this study is to compare the effect of two non-invasive neuromodulation targets in patients meeting WHO criteria for the post-COVID condition. A randomized, parallel, double-blind study will be conducted. Patients will receive 15 neuromodulation sessions through transcranial electrical stimulation for 3 weeks, associated with cognitive stimulation during therapy. The main objective will be to evaluate the change in physical fatigue. As secondary objectives, changes in cognition, depression, pain, quality of sleep and quality of life will be evaluated. The objective of this study is to evaluate the effect of two targets (left dorsolateral prefrontal and M1) of the neuromodulation intervention, together with cognitive stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COVID-19 at least 6 months before the participation in the study.
* Diagnosis of post-COVID condition according to WHO criteria.
* Age 18-65 years.
* Spanish as native language.
* Sign of written informed consent.

Exclusion Criteria:

* History of stroke
* History of traumatic brain injury or central nervous system infection
* Diagnosis of other neurological or medical disorder that could impact on fatigue.
* Diagnosis of active psychiatric disorder potentially impacting on fatigue or cognitive function.
* Chemotherapy or radiotherapy for cancer.
* Severe sensory deficits (e.g. visual loss) that could limit assessments included int the study protocol.
* Taking drugs or uncontrolled medical disorder potentially causing or worsening fatigue. Specifically, uncontrolled adrenal insufficiency, miastenic syndromes, thyroid disorders, cardiac failure, chronic kidney disorders and neurodegenerative disorders are excluded.
* History of abuse of alcohol or other toxics.
* Any contraindication for transcranial electric stimulation: epilepsy, pregnancy, metallic implants, brain devices, pacemakers, head injuries).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale (score) | 1 month
  Physical fatigue

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) (score) | 1 month
  Physical and cognitive fatigue
FLEI scale (score) | 1 month
  Subjective cognition.
Beck Depression Inventory (2nd version) (score) | 1 month
  Depressive symptoms
Pittsburgh Sleep Quality Index (score) | 1 month
  Sleep quality
Brief Pain Inventory (score) | 1 month
  Pain

CONTACTS AND LOCATIONS:
Overall Officials: Jordi A Matias-Guiu, PhD, Principal Investigator — Hospital Clinico San Carlos
Locations (1):
- Hospital Clínico San Carlos., Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the end of the study and publication of the results. For 5 years.
Access Criteria: Data will be shared after reasonable request to the principal investigator.

REFERENCES:
- [Derived] Oliver-Mas S, Matias-Guiu JA, Delgado-Alonso C, Gil-Martinez L, Cuevas C, Polidura C, Fernandez-Romero L, Matias-Guiu A, Gomez-Ruiz N, Gil-Moreno MJ, Yus-Fuertes M, Matias-Guiu J, Diez-Cirarda M. A randomized comparative feasibility study of neuromodulation and cognitive training for post-COVID fatigue. Sci Rep. 2025 Jul 23;15(1):26818. doi: 10.1038/s41598-025-09772-8. PMID 40702022